CLINICAL TRIAL: NCT03154502
Title: Sodium Urinary Excretion Measurement in Ecuadorian Population
Brief Title: Sodium Intake in Ecuadorian Population
Status: Completed | Type: Observational
Sponsor: Universidad San Francisco de Quito (Other)
Responsible Party: Principal Investigator, Ivan Sisa, Associate Professor, Universidad San Francisco de Quito
Other Study IDs: HUBI-1022
Record Dates: First submitted 2017-05-12; First posted 2017-05-16 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Dietary Habits; Risk Factor, Cardiovascular; Nutritional Disorder
Keywords: Sodium intake; Urinary sodium excretion
MeSH Terms: conditions — Feeding Behavior; Nutrition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Urinary sodium excretion — Urinary sodium and potassium were measured using the Ion-Selective Electrode (ISE) indirect Na-K-Cl for Gen.2 (Roche Diagnostic, Switzerland).

SUMMARY:
This study is aim to determine the sodium intake in Ecuadorian population that is an unknown information at present. For that, 24h urine samples will be collected from 130 subjects working either at tue USFQ or HDLV to measure sodium excretion.

ELIGIBILITY:
Inclusion Criteria:

* None

Exclusion Criteria:

* unable to provide informed consent
* unable to provide 24-hr urine excretion sample
* those with a known history of heart or kidney failure, stroke, and liver disease
* those using diuretics, multivitamins, NSADs, or prostaglandins during the last two weeks
* pregnant women

Ages: 25 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Will be enrolled a sample of 178 adults aged 25 to 64 years. The research team, who have faculty appointments in USFQ, supervised the collection of the urine samples. We invited a broad spectrum of employees (which included health care workers, professors, and custodial staff) from both institutions to participate in the study.
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2016-10-30 (Actual); Study Completion 2016-10-30 (Actual)

PRIMARY OUTCOMES:
Urinary sodium excretion | 1 year
  Amount of sodium in 24h urine collection

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Teran, MD, PhD, Study Director — Universidad San Francisco de Quito

IPD SHARING:
Plan to Share IPD: No